CLINICAL TRIAL: NCT07061977
Title: NRG-GY037: A Phase III Study of Induction Pembrolizumab and Chemotherapy Followed by Chemoradiation and Pembrolizumab Versus Chemoradiation and Pembrolizumab Both Followed by Pembrolizumab for High Risk Locally Advanced Cervical Cancer
Brief Title: Induction Pembrolizumab and Chemotherapy Followed by Pembrolizumab Before Chemoradiation and Pembrolizumab Maintenance Compared to Standard Chemoradiation With Pembrolizumab Followed by Pembrolizumab Maintenance in High-Risk Cervical Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-04695; NCI-2025-04695 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY037 (Other: NRG Oncology); NRG-GY037 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Cervical Adenocarcinoma; Locally Advanced Cervical Adenosquamous Carcinoma; Locally Advanced Cervical Squamous Cell Carcinoma; Stage IIIA Cervical Cancer FIGO 2018; Stage IIIB Cervical Cancer FIGO 2018; Stage IIIC1 Cervical Cancer FIGO 2018; Stage IIIC2 Cervical Cancer FIGO 2018; Stage IVA Cervical Cancer FIGO 2018
MeSH Terms: interventions — Specimen Handling; Brachytherapy; Carboplatin; X-Rays; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Congresses as Topic; Radiation; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Standard care) (Active Comparator): CHEMORADIATION: Patients receive cisplatin IV QW for 5 weeks and pembrolizumab IV over 30 minutes Q3W for 5 doses. Patients also undergo radiation therapy with EBRT or IMRT once daily 5 days per week for 25-29 treatments in weeks 1-5 followed by brachytherapy up to twice per week for 4-5 treatments in weeks 5-7. Treatment is given in the absence of disease progression or unacceptable toxicity
  MAINTENANCE: Patients receive pembrolizumab IV over 30 minutes Q6W for 14 cycles in the absence of disease progression or unacceptable toxicity.
  Patients undergo PET scan, CT scan, chest x-ray and/or MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Radiation: Brachytherapy; Procedure: Chest Radiography; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography
- Arm 2 (induction and standard care) (Experimental): INDUCTION: Patients receive carboplatin IV and paclitaxel IV QW on weeks 1-3 and pembrolizumab IV over 30 minutes Q3W on week 1 for each cycle. Cycles repeat every 3 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity.
  CHEMORADIATION: Patients receive cisplatin IV QW for 5 weeks and pembrolizumab IV over 30 minutes every Q3W for 5 doses. Patients also undergo radiation therapy with EBRT or IMRT once daily 5 days per week for 25-29 treatments in weeks 7-11 followed by brachytherapy up to twice per week for 4-5 treatments in weeks 11-13. Treatment is given in the absence of disease progression or unacceptable toxicity
  MAINTENANCE: Patients receive pembrolizumab IV over 30 minutes Q6W for 14 cycles in the absence of disease progression or unacceptable toxicity.
  Patients undergo PET scan, CT scan, chest x-ray and/or MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Radiation: Brachytherapy; Drug: Carboplatin; Procedure: Chest Radiography; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Biological: Pembrolizumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Radiation: Brachytherapy — Undergo brachytherapy
  Other Names: Brachytherapy, NOS; Internal Radiation; Internal Radiation Brachytherapy; Internal Radiation Therapy; Radiation Brachytherapy; Radiation, Internal
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm 2 (induction and standard care)
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm 2 (induction and standard care)
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase III trial compares the addition of induction chemotherapy, with carboplatin, paclitaxel and pembrolizumab, to chemotherapy and radiation, with cisplatin and pembrolizumab followed by pembrolizumab maintenance for the treatment of patients with cervical cancer that has spread to nearby tissue or lymph nodes (locally advanced). Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of cancer cells. Paclitaxel is in a class of medications called antimicrotubule agents. It stops cancer cells from growing and dividing and may kill them. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of cancer cells. Adding induction chemotherapy to the usual treatment of chemotherapy and radiation followed by maintenance may be more effective in treating patients with high risk, locally advanced cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether induction immunotherapy (IO) and chemotherapy prior to concurrent chemoradiation therapy (CCRT) + IO improves progression-free survival (PFS) compared to CCRT+IO alone.

SECONDARY OBJECTIVES:

I. To assess whether induction IO and chemotherapy prior to CCRT+IO improves the overall survival (OS) compared to CCRT+IO alone.

II. To determine the nature and degree of toxicity of induction IO and chemotherapy prior to CCRT + IO as compared to concurrent CCRT+IO as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

III. To determine the impact on CCRT start, CCRT completion time, and number of cycles of cisplatin administered; with induction IO and chemotherapy prior to CCRT+IO arm as compared to CCRT+IO.

IV. To assess the association between allostatic load and PFS/OS. V. To assess the predictive value of the integrated biomarker: PD-L1 expression at baseline for progression free survival.

VI. To assess the prognostic and predictive value of the integrated biomarker: circulating tumor deoxyribonucleic acid (ctDNA) at baseline and at 3 months post radiation therapy (RT) for progression free survival.

VII. To explore radiotherapy quality pretreatment scores conducted by expert review with assistance from artificial intelligence (AI) models and correlation with outcomes.

EXPLORATORY OBJECTIVES:

I. To assess the evolution of T cell receptor (TCR) repertoire on treatment and its correlation with clinical outcomes.

II. To identify pre-treatment tumor microenvironment biomarkers predictive of outcomes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1:

CHEMORADIATION: Patients receive cisplatin intravenously (IV) once weekly (QW) for 5 weeks and pembrolizumab IV over 30 minutes every 3 weeks (Q3W) for 5 doses. Patients also undergo radiation therapy once daily 5 days per week for 25-29 treatments in weeks 1-5 followed by brachytherapy up to twice per week for 4-5 treatments in weeks 5-7. Treatment is given in the absence of disease progression or unacceptable toxicity

MAINTENANCE: Patients receive pembrolizumab IV over 30 minutes every 6 weeks (Q6W) for 15 cycles in the absence of disease progression or unacceptable toxicity.

Patients undergo positron emission tomography (PET) scan, computed tomography (CT) scan, chest x-ray and/or magnetic resonance imaging (MRI) and blood sample collection throughout the study.

ARM 2:

INDUCTION: Patients receive carboplatin IV and paclitaxel IV QW on weeks 1-3 and pembrolizumab IV over 30 minutes Q3W on weeks 1 for each cycle. Cycles repeat every 3 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity.

CHEMORADIATION: Patients receive cisplatin IV QW for 5 weeks and pembrolizumab IV over 30 minutes every Q3W for 5 doses. Patients also undergo radiation therapy once daily 5 days per week for 25-29 treatments in weeks 7-11 followed by brachytherapy up to twice per week for 4-5 treatments in weeks 11-13. Treatment is given in the absence of disease progression or unacceptable toxicity

MAINTENANCE: Patients receive pembrolizumab IV over 30 minutes Q6W for 14 cycles in the absence of disease progression or unacceptable toxicity.

Patients undergo PET scan, CT scan, chest x-ray and/or MRI and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed newly diagnosed cervical cancer. Eligible pathologic types: squamous cell carcinoma, adenocarcinoma, adenosquamous cell carcinoma
* Patients must have locally advanced cervical cancer (LACC) with T3 or T4 disease with or without lymph node involvement:

  * IIIA (T3aN0M0)
  * IIIB (T3bN0M0)
  * IIIC1(T3aN1M0, T3bN1M0)
  * IIIC2 (T3aN2M0, T3bN2M0)
  * IVA (T4aN0M0, T4aN1M0, T4aN2M0) No prior hysterectomy defined as removal of the entire uterus.
  * NOTE: prior partial/subtotal hysterectomy for reasons other than cervical cancer are eligible to participate in the study. No plan to perform a hysterectomy as part of initial cervical cancer therapy.

No paraaortic lymph node (PALN) metastases above the T12/L1 interspace.

* Note: Nodal status can be confirmed by imaging (CT, MRI, or PET/CT), fine needle aspirate/core biopsy, extra peritoneal biopsy, laparoscopic biopsy, or lymphadenectomy.

Radiologic definition of lymph node staging:

* N1:

  * One or more pelvic lymph nodes with short axis diameter of ≥ 15 mm (axial plane) by CT or MRI, and/or
  * One or more pelvic lymph nodes with short axis diameter of ≥ 10 mm and standardized uptake value maximum (SUVmax) ≥ 2.5 by fludeoxyglucose (FDG)-PET
* N2:

  * One or more para-aortic lymph node with short axis diameter of ≥ 15 mm (axial plane) by CT or MRI, and/or
  * One or more para-aortic lymph node with short axis diameter of ≥ 10 mm and SUVmax ≥ 2.5 by FDG-PET

    * No prior definitive surgical, radiation, or systemic therapy for cervical cancer
    * No prior immunotherapy
    * No prior pelvic radiation therapy for any disease
    * Age ≥ 18
    * Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
    * Not pregnant and not nursing
    * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
    * Platelets ≥ 100,000 cells/mm^3
    * Hemoglobin ≥ 8 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobulin [Hgb] ≥ 8 g/dl is acceptable)
    * Creatinine clearance (CrCL) of ≥ 50 mL/min by the Cockcroft-Gault formula
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (patients with known Gilbert's disease who have bilirubin level ≤ 3 x institutional ULN may be enrolled)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x institutional ULN
    * Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
    * No active infection requiring parenteral antibiotics
    * No live vaccine within 30 days prior to registration. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacille Calmette Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed
    * No diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior registration
    * No active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
    * No history of (non-infectious) pneumonitis that required steroids, or current pneumonitis
    * No history of allergic reaction to the study agent(s) or compounds of similar chemical or biologic composition to the study agent(s) (or any of its excipients)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From randomization to time of progression or death from any cause, whichever occurs first, or date of last contact if neither progression nor death has occurred, up to 7 years
  Analysis will be performed using a one-sided log-rank test stratified by factors declared at randomization when (at least) 190 PFS events are observed in both arms. Patients will be grouped by their randomized treatment for intention-to-treat (ITT) analyses, supported by patients in ITT population. Treatment hazard ratio and confidence will be estimated using Cox proportional hazard models specified with a main effect for the randomized treatment assignment and stratified by factors declared at randomization. PFS at 2 years will be estimated using Kaplan-Meier method for each arm.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, up to 7 years
  The OS treatment hypothesis test (Arm 2 versus [vs.] Arm 1) will be based on a 1-sided log-rank test, stratified by the factors specified at randomization. Comparisons of the OS distributions by treatment arm will be described using Kaplan-Meier methods. Treatment hazard ratio estimates and their 95% confidence intervals will be estimated using a multivariable proportional hazards model specified with main effects for the randomized treatment assignment (Arm 2 vs Arm 1) and stratified by the factors declared at randomization.
Incidence of adverse events (AEs) | Up to 7 years
  Assessed by Common Terminology Criteria for Adverse Events version 5.0. The nature, frequency, and degree of toxicity will be tabulated at the System Organ Class and AE-specific term levels. Tabulations will show the number and percentage of patients by maximum grade, within the treatment group received, regardless of the randomized treatment assignment. Differences in the level of toxicities by treatment arm will be assessed by classifying them as severe (grade 3 or higher) or not severe (grade 2 or lower) and examining the relative proportion of severe toxicities by Fisher's exact test.
Duration of concurrent chemoradiation therapy (CCRT) completion | From CCRT start date to CCRT end date
  Will be summarized and compared using 2-sample Wilcoxon rank sum tests. The proportion of patients with a delayed time to initiate CCRT by 2 weeks or more will be estimated and investigated by Fisher's exact test.
Number of cycles of cisplatin | From 7 days after the last dose of induction chemotherapy to the CCRT start date for Arm 2, the planned CCRT start date to actual CCRT start date for Arm 1
  Will be summarized and compared using 2-sample Wilcoxon rank sum tests.
Allostatic load | Up to 2 years
  Will be summarized by treatment arm, and its association with OS will be evaluated using Cox PH model adjusted with main effects for the randomized treatment assignment (Arm 2 vs Arm 1) and stratified by the factors declared at randomization.
Tumor PD-L1 expression | At baseline
  The predictive value of tumor PD-L1 expression at baseline for PFS will be investigated using Cox PH model adjusted with main effects for the randomized treatment assignment (Arm 2 vs Arm 1) and stratified by the factors declared at randomization.
Circulating tumor deoxyribonucleic acid expression | At baseline and at 3 months post radiation therapy
  Will be summarized by treatment arm and by collection time. Will be investigated using Cox PH model adjusted with main effects for the randomized treatment assignment (Arm 2 vs Arm 1) and stratified by the factors declared at randomization.
Radiation quality pre-treatment score | At time of radiation
  Will be summarized by treatment arm, and its associations with PFS and OS will be evaluated using Cox PH model adjusted with main effects for the randomized treatment assignment (Arm 2 vs Arm 1) and stratified by the factors declared at randomization.

OTHER OUTCOMES:
T cell receptor (TCR) expression | Up to 7 years
  Will be summarized by treatment arm, and its correlation with PFS/OS will be investigated using Cox PH model adjusted with main effects for the randomized treatment assignment (Arm 2 vs Arm 1) and stratified by the factors declared at randomization. Repeated measure methods (e.g., linear mixed model) will be used for exploration of TCR evolution/trajectory on treatment.
Tumor microenvironment | At baseline
  The predictive values of each of the pre-treatment tumor microenvironment biomarkers for PFS and OS will be investigated using Cox PH model adjusted with main effects for the randomized treatment assignment (Arm 2 vs Arm 1) and stratified by the factors declared at randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti S Mayadev, Principal Investigator — NRG Oncology
Locations (121):
- United States (121):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope Upland, Upland, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Northwell Health Physicians Partners Radiation Medicine at Queens, Forest Hills, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Upstate Cancer Center Radiation Oncology at Oswego, Oswego, New York
  - Queens Cancer Center, Rego Park, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Upstate Cancer Center at Hill Radiation Oncology, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Duke University Medical Center, Durham, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Saint Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm